CLINICAL TRIAL: NCT04730557
Title: Reducing Obesity and Cartilage Compression in Knees
Acronym: ROCCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00102409
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Obesity; Osteoarthritis; Knee Osteoarthritis
Keywords: Weight Loss; MRI; Arthritis; Knee Health
MeSH Terms: conditions — Obesity; Osteoarthritis; Osteoarthritis, Knee; Weight Loss; Arthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight-Loss (Experimental): Participants in the weight-loss intervention arm of the study will be enrolled in an individualized 6-month intervention designed to achieve a 10% reduction of body weight relative to baseline. Each participant receives a calorie (kcal) prescription derived from calculations of estimated total energy expenditure (TEE) based on weight, height, sex, age, and activity level using equations developed by the Institute of Medicine [29]. Prescribed kcal levels are adjusted downward from the TEE to achieve a weekly weight loss of 1 to 2 pounds, generally a deficit of 500-1000 kcal/day. Intervention activities include individual diet counseling, group support, goal setting, self-monitoring, stress management, and problem solving. Weekly group support and education sessions, along with daily food journaling and weekly weigh-ins, are recognized approaches for successful weight loss [30-32]. Once the weight loss goal is achieved, diets will be liberalized for weight maintenance.
  Interventions: Behavioral: Weight Loss
- Wellness Education (No Intervention): Control participants will be counseled to maintain their baseline body weight and level of physical activity. They will report weights weekly and if their weight deviates from baseline they will be asked to keep daily food logs and counseled to return calorie intakes to weight maintenance level. To document diet intakes/adherence, 3-day food records will be collected at months 0, 3, and 6 and analyzed for calorie and nutrient composition. Participants will be encouraged not to change their physical activity levels from baseline and their activity will be monitored by Actigraph activity monitors worn in 7-day periods at months 0, 3, and 6. In addition, each participant will be invited to enter the weight loss intervention after completion of the health education control course.

INTERVENTIONS:
Behavioral: Weight Loss — Each participant receives a calorie (kcal) prescription derived from calculations of estimated total energy expenditure (TEE) based on weight, height, sex, age, and activity level using equations developed by the Institute of Medicine [29]. Prescribed kcal levels are adjusted downward from the TEE to achieve a weekly weight loss of 1 to 2 pounds, generally a deficit of 500-1000 kcal/day. Weekly intervention sessions and activities will be delivered virtually using Microsoft Teams, Duke ZOOM or Duke Webex and led by Registered Dietitians.
  Arms: Weight-Loss

SUMMARY:
OA is a degenerative joint disease that involves the degradation of articular cartilage and underlying subchondral bone. Obesity is identified as a critical and potentially modifiable risk factor for the development and progression of OA. The first objective of the study is to determine the effects of obesity on cartilage composition and function. The second objective of the study is to determine whether weight loss restores cartilage composition and function. Study activities would require getting MR Imaging, evaluation of joint loading using gait analysis techniques, cartilage strain measurement, and participating in weight loss intervention. The study will target a population age group between 18 and 45 years with a BMI greater than or equal to 29. Data analyses will be blinded to reduce potential bias. All subjects participating in this study will be informed of the risks involved and sign an IRB-approved consent form.

DETAILED DESCRIPTION:
Appropriate study power will be achieved with 35 participants in the weight loss group and 35 participants in the weight maintenance control group (see Data Analysis and Statistical Considerations). We will recruit and enroll obese (BMI ≥29 - ≤40) men and women, age 18 to 45, with no previous history of lower extremity injury, no evidence of symptoms OA, no knee misalignment (neutral alignment between 178° and 182°), or other injury that would prevent them from performing the walking task required by this study. All inclusion criteria specific to knee injury, OA, and alignment will be verified by MRI scan. All participants in this study will be informed of the risks involved. Upon expressing interest in study participation, participants will be asked questions to determine whether they are free of lower extremity injury and their height and weight will also be recorded to determine their BMI. Potential participants will be pre-screened by phone using a phone script with a list of questions. Once it is determined they meet all study inclusion criteria, they will be invited to attend a consent meeting.

ELIGIBILITY:
Inclusion Criteria:

* BMI (BMI ≥29 - <40)
* Age between 18 - 45

Exclusion Criteria:

* History of lower extremity injury
* Evidence of symptoms of knee OA
* Knee misalignment
* Evidence of pregnancy
* Thigh unable to fit in MRI coil
* Body waist fit in MRI
* Have no metals in the body

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cartilage strain/thickness at 3 and 6 months | Baseline, 3 months, and 6 months
  We will use MRI to detect change in cartilage strain/thickness at 3 and 6 months

SECONDARY OUTCOMES:
Change from baseline in cartilage composition at 3 and 6 months | Baseline, 3 months, and 6 months
  We will use MRI to detect change in cartilage composition at 3 and 6 months
Change from baseline in inflammation at 3 and 6 months | Baseline, 3 months, and 6 months
  Serum and urine biomarkers will be collected to determine levels of inflammation.
Change from baseline in cartilage degeneration at 3 and 6 months | Baseline, 3 months, and 6 months
  We will use serum biomarkers to determine cartilage degeneration
Change from baseline in biomarkers of insulin resistance and beta-cell function at 3 and 6 months | Baseline, 3 months, and 6 months
  We will use serum biomarkers to determine insulin resistance and beta-cell function
Change from baseline in muscle strength at 3 and 6 months | Baseline, 3 months, and 6 months
  Isokinetic dynamometer will be used to determine peak torque of knee extensor and flexor
Change from baseline in body weight at 3 and 6 months | Baseline, 3 months, and 6 months
  Body weight as measured by Bodpod
Change from baseline in fat mass (kg) at 3 and 6 months | Baseline, 3 months, and 6 months
  Body fat mass (kg) as measured by Bodpod
Change from baseline in fat mass (%) at 3 and 6 months | Baseline, 3 months, and 6 months
  Body fat mass (%) as measured by Bodpod
Change from baseline in lean mass (%) at 3 and 6 months | Baseline, 3 months, and 6 months
  Body lean mass (%) as measured by Bodpod
Change from baseline in lean mass (kg) at 3 and 6 months | Baseline, 3 months, and 6 months
  Body lean mass (%) as measured by Bodpod
Change from baseline in 6-minute walk (meters) at 3 and 6 months | Baseline, 3 months, and 6 months
  Distanced (meters) walked in 6 minutes
Change from baseline in umbilical waist circumference at 3 and 6 months | Baseline, 3 months, and 6 months
  Body proportions will be measured at the umbilical waist using a Gulick II tape measure with the tape placed directly on the skin (not over clothes). Measurement will be taken once at each location before completing a second measurement, and an average of the two will be recorded. A third measurement will be taken if the first two measurements are >0.5 cm.
Change from baseline in minimal waist circumference at 3 and 6 months | Baseline, 3 months, and 6 months
  Body proportions will be measured at the minimal waist using a Gulick II tape measure with the tape placed directly on the skin (not over clothes). Measurement will be taken once at each location before completing a second measurement, and an average of the two will be recorded. A third measurement will be taken if the first two measurements are >0.5 cm.
Change from baseline in hip circumference at 3 and 6 months | Baseline, 3 months, and 6 months
  Body proportions will be measured at the hip circumference using a Gulick II tape measure with the tape placed directly on the skin (not over clothes). Measurement will be taken once at each location before completing a second measurement, and an average of the two will be recorded. A third measurement will be taken if the first two measurements are >0.5 cm.
Change from baseline total calories at 3 and 6 months | Baseline, 3 months, and 6 months
  Total calories will be measured using a 3-day food record (participant records everything they eat and drink for three days)
Change from baseline macronutrients at 3 and 6 months | Baseline, 3 months, and 6 months
  Total calories will be measured using a 3-day food record (participant records everything they eat and drink for three days)
Change in activity (intensity levels) at 3 and 6 months | Baseline, 3 months, and 6 months
  Activity intensity levels using an actigraphy device worn for 7 days at each time point
Change in steps at 3 and 6 months | Baseline, 3 months, and 6 months
  Steps will be determined using an actigraphy device worn for 7 days at each time point
Change in Healthy Eating Index at 3 months and 6 months | Baseline, 3 months, and 6 months
  Healthy Eating Index (HEI-2015) calculated from Dietary History Questionnaire III (DHQIII, National Cancer Institute) at each time point. The HEI score ranges from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Americans..

CONTACTS AND LOCATIONS:
Overall Officials: Lou DeFrate, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Pereira D, Peleteiro B, Araujo J, Branco J, Santos RA, Ramos E. The effect of osteoarthritis definition on prevalence and incidence estimates: a systematic review. Osteoarthritis Cartilage. 2011 Nov;19(11):1270-85. doi: 10.1016/j.joca.2011.08.009. Epub 2011 Aug 24. PMID 21907813
- [Background] Kopec JA, Rahman MM, Berthelot JM, Le Petit C, Aghajanian J, Sayre EC, Cibere J, Anis AH, Badley EM. Descriptive epidemiology of osteoarthritis in British Columbia, Canada. J Rheumatol. 2007 Feb;34(2):386-93. Epub 2006 Dec 15. PMID 17183616
- [Background] Goldring SR, Goldring MB. Bone and cartilage in osteoarthritis: is what's best for one good or bad for the other? Arthritis Res Ther. 2010;12(5):143. doi: 10.1186/ar3135. Epub 2010 Oct 19. PMID 21044355
- [Background] Day JS, Ding M, van der Linden JC, Hvid I, Sumner DR, Weinans H. A decreased subchondral trabecular bone tissue elastic modulus is associated with pre-arthritic cartilage damage. J Orthop Res. 2001 Sep;19(5):914-8. doi: 10.1016/S0736-0266(01)00012-2. PMID 11562141
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, part I: critical appraisal of existing treatment guidelines and systematic review of current research evidence. Osteoarthritis Cartilage. 2007 Sep;15(9):981-1000. doi: 10.1016/j.joca.2007.06.014. Epub 2007 Aug 27. PMID 17719803
- [Background] Ringdahl E, Pandit S. Treatment of knee osteoarthritis. Am Fam Physician. 2011 Jun 1;83(11):1287-92. PMID 21661710
- [Background] Kretzer JP, Jakubowitz E, Sonntag R, Hofmann K, Heisel C, Thomsen M. Effect of joint laxity on polyethylene wear in total knee replacement. J Biomech. 2010 Apr 19;43(6):1092-6. doi: 10.1016/j.jbiomech.2009.12.016. Epub 2010 Jan 13. PMID 20074735
- [Background] Lahuec C, Almouahed S, Arzel M, Gupta D, Hamitouche C, Jezequel M, Stindel E, Roux C. A self-powered telemetry system to estimate the postoperative instability of a knee implant. IEEE Trans Biomed Eng. 2011 Mar;58(3):822-5. doi: 10.1109/TBME.2010.2069099. Epub 2010 Aug 30. PMID 20805049
- [Background] Felson DT. Relation of obesity and of vocational and avocational risk factors to osteoarthritis. J Rheumatol. 2005 Jun;32(6):1133-5. No abstract available. PMID 15977343
- [Background] Griffin TM, Guilak F. Why is obesity associated with osteoarthritis? Insights from mouse models of obesity. Biorheology. 2008;45(3-4):387-98. PMID 18836239
- [Background] Browning RC, Kram R. Effects of obesity on the biomechanics of walking at different speeds. Med Sci Sports Exerc. 2007 Sep;39(9):1632-41. doi: 10.1249/mss.0b013e318076b54b. PMID 17805097
- [Background] Englund M, Lohmander LS. Risk factors for symptomatic knee osteoarthritis fifteen to twenty-two years after meniscectomy. Arthritis Rheum. 2004 Sep;50(9):2811-9. doi: 10.1002/art.20489. PMID 15457449
- [Background] Felson DT. Does excess weight cause osteoarthritis and, if so, why? Ann Rheum Dis. 1996 Sep;55(9):668-70. doi: 10.1136/ard.55.9.668. No abstract available. PMID 8882146
- [Background] Felson DT. Weight and osteoarthritis. Am J Clin Nutr. 1996 Mar;63(3 Suppl):430S-432S. doi: 10.1093/ajcn/63.3.430. PMID 8615335
- [Background] Murphy L, Schwartz TA, Helmick CG, Renner JB, Tudor G, Koch G, Dragomir A, Kalsbeek WD, Luta G, Jordan JM. Lifetime risk of symptomatic knee osteoarthritis. Arthritis Rheum. 2008 Sep 15;59(9):1207-13. doi: 10.1002/art.24021. PMID 18759314
- [Background] Grotle M, Hagen KB, Natvig B, Dahl FA, Kvien TK. Obesity and osteoarthritis in knee, hip and/or hand: an epidemiological study in the general population with 10 years follow-up. BMC Musculoskelet Disord. 2008 Oct 2;9:132. doi: 10.1186/1471-2474-9-132. PMID 18831740
- [Background] Carman WJ, Sowers M, Hawthorne VM, Weissfeld LA. Obesity as a risk factor for osteoarthritis of the hand and wrist: a prospective study. Am J Epidemiol. 1994 Jan 15;139(2):119-29. doi: 10.1093/oxfordjournals.aje.a116974. PMID 8296779
- [Background] Oliveria SA, Felson DT, Cirillo PA, Reed JI, Walker AM. Body weight, body mass index, and incident symptomatic osteoarthritis of the hand, hip, and knee. Epidemiology. 1999 Mar;10(2):161-6. PMID 10069252
- [Background] Messier SP, Loeser RF, Miller GD, Morgan TM, Rejeski WJ, Sevick MA, Ettinger WH Jr, Pahor M, Williamson JD. Exercise and dietary weight loss in overweight and obese older adults with knee osteoarthritis: the Arthritis, Diet, and Activity Promotion Trial. Arthritis Rheum. 2004 May;50(5):1501-10. doi: 10.1002/art.20256. PMID 15146420
- [Background] Serebrakian AT, Poulos T, Liebl H, Joseph GB, Lai A, Nevitt MC, Lynch JA, McCulloch CE, Link TM. Weight loss over 48 months is associated with reduced progression of cartilage T2 relaxation time values: data from the osteoarthritis initiative. J Magn Reson Imaging. 2015 May;41(5):1272-1280. doi: 10.1002/jmri.24630. Epub 2014 Apr 4. PMID 24700497
- [Background] Felson DT, Zhang Y, Anthony JM, Naimark A, Anderson JJ. Weight loss reduces the risk for symptomatic knee osteoarthritis in women. The Framingham Study. Ann Intern Med. 1992 Apr 1;116(7):535-9. doi: 10.7326/0003-4819-116-7-535. PMID 1543306
- [Background] Abu-Abeid S, Wishnitzer N, Szold A, Liebergall M, Manor O. The influence of surgically-induced weight loss on the knee joint. Obes Surg. 2005 Nov-Dec;15(10):1437-42. doi: 10.1381/096089205774859281. PMID 16354524
- [Background] Powell A, Teichtahl AJ, Wluka AE, Cicuttini FM. Obesity: a preventable risk factor for large joint osteoarthritis which may act through biomechanical factors. Br J Sports Med. 2005 Jan;39(1):4-5. doi: 10.1136/bjsm.2004.011841. PMID 15618330
- [Background] Aspden RM. Obesity punches above its weight in osteoarthritis. Nat Rev Rheumatol. 2011 Jan;7(1):65-8. doi: 10.1038/nrrheum.2010.123. Epub 2010 Aug 17. PMID 20717100
- [Background] Messier SP, Gutekunst DJ, Davis C, DeVita P. Weight loss reduces knee-joint loads in overweight and obese older adults with knee osteoarthritis. Arthritis Rheum. 2005 Jul;52(7):2026-32. doi: 10.1002/art.21139. PMID 15986358
- [Background] Messier SP, Mihalko SL, Legault C, Miller GD, Nicklas BJ, DeVita P, Beavers DP, Hunter DJ, Lyles MF, Eckstein F, Williamson JD, Carr JJ, Guermazi A, Loeser RF. Effects of intensive diet and exercise on knee joint loads, inflammation, and clinical outcomes among overweight and obese adults with knee osteoarthritis: the IDEA randomized clinical trial. JAMA. 2013 Sep 25;310(12):1263-73. doi: 10.1001/jama.2013.277669. PMID 24065013
- [Background] Trumbo P, Schlicker S, Yates AA, Poos M; Food and Nutrition Board of the Institute of Medicine, The National Academies. Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids. J Am Diet Assoc. 2002 Nov;102(11):1621-30. doi: 10.1016/s0002-8223(02)90346-9. No abstract available. PMID 12449285
- [Background] Seagle HM, Strain GW, Makris A, Reeves RS; American Dietetic Association. Position of the American Dietetic Association: weight management. J Am Diet Assoc. 2009 Feb;109(2):330-46. doi: 10.1016/j.jada.2008.11.041. PMID 19244669
- [Background] Hollis JF, Gullion CM, Stevens VJ, Brantley PJ, Appel LJ, Ard JD, Champagne CM, Dalcin A, Erlinger TP, Funk K, Laferriere D, Lin PH, Loria CM, Samuel-Hodge C, Vollmer WM, Svetkey LP; Weight Loss Maintenance Trial Research Group. Weight loss during the intensive intervention phase of the weight-loss maintenance trial. Am J Prev Med. 2008 Aug;35(2):118-26. doi: 10.1016/j.amepre.2008.04.013. PMID 18617080
- [Background] Streit KJ, Stevens NH, Stevens VJ, Rossner J. Food records: a predictor and modifier of weight change in a long-term weight loss program. J Am Diet Assoc. 1991 Feb;91(2):213-6. PMID 1991935